CLINICAL TRIAL: NCT07034417
Title: Investigation The Effectiveness Of Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı - BETY) In Individuals With Fibromyalgia
Brief Title: The Effectiveness Of BETY In Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aysima Barlak (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other); Alanya Alaaddin Keykubat University Alanya Training and Research Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Aysima Barlak, PT, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 03-03
Record Dates: First submitted 2025-03-18; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia
Keywords: biopsychosocial model; pain; functional capacity; depression; anxiety; quality of life
MeSH Terms: conditions — Fibromyalgia; Pain; Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı - BETY)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BETY Group (Experimental): BETY exercise sessions
  Interventions: Other: Exercise
- Control Group (Other): Home exercise program
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Exercise — Cognitive Exercise Therapy Approach
  Arms: BETY Group
Other: Home exercise — Home exercise
  Arms: Control Group

SUMMARY:
Fibromyalgia Syndrome (FMS) is a nonarticular, chronic rheumatic disorder of unknown etiology characterized by widespread musculoskeletal pain, impaired sleep quality, fatigue and the presence of identified tender points. Pain, the main symptom of the disease, is described as chronic and widespread. It is reported that the pain usually starts in the neck and shoulders but becomes widespread by being felt in various parts of the body during the day. Although it is difficult to localize the pain, it is reported to be localized to the paracervical and trapezius muscle and paralumbar and gluteal body parts.

Cognitive Exercise Therapy Approach is an innovative exercise approach developed on the basis of biopsychosocial model on individuals with rheumatism. This method has a unique scale that offers biopsychosocial assessment. There is the Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ). Validity, reliability and sensitivity studies of BETY-BQ have been conducted in individuals with fibromyalgia. This study aims to examine the effect of BETY, an exercise approach developed on the basis of the biopsychosocial model, on individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia
* 18 years of age or older
* Being literate
* Having read and signed the informed consent
* Not exercising regularly in the last 3 months

Exclusion Criteria:

* Having a malignant disease
* Pregnancy
* Having chronic infectious or other rheumatologic diseases
* Having undergone a surgical operation in the last 6 months
* Collagen tissue disease
* History of peripheral vascular disease or neuropathy
* Presence of diseases that cannot be controlled and prevent exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-12 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach (BETY)- Biopsychosocial Questionnaire | 3 mounths
  The BETY Questionnaire was developed on rheumatic patients and was introduced to the literature as a standardized biopsychosocial measurement tool as a result of improving the definitions of recovery from patients with expert opinions and statistical analysis. Scoring of the scale is done using a 5-point Likert system, each item is scored between 0 and 4 points, and a high total score in the scale consisting of a total of 30 items indicates a high biopsychosocial impact.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale (HADS) | 3 mounths
  Although the HADS was developed 20 years ago for the clinical measurement of anxiety and depression levels and was originally developed for hospitalized individuals, it now has a wide spectrum of use and can be used in many situations, including healthy people. Seven of the 14 items provide insight into the level of anxiety, while seven include questions about the level of depression. Each question is scored between 0 and 3, with a high score indicating high affectivity. Anxiety and depression sub-parameters are scored separately and 11 points and above are considered abnormal.
Health Asessement Questionnaire (HAQ) | 3 mounths
  It is a scale developed in individuals with rheumatoid arthritis and can be used in a wide range of populations while assessing all rheumatic disease groups. It has 8 subheadings and consists of a total of 20 questions. Sub-headings include dressing, sitting and staying, eating, walking, hygiene, reaching, grasping and activities of daily living. Each answer is scored between 0 and 3 points and the higher the score, the more difficult the activity is.
Short Form - 36 | 3 mounths
  SF-36 scale will be used to determine the level of health status and quality of life of individuals.SF-36 is a patient-oriented assessment scale created in the United States of America that allows for general health screening.Each sub-parameter is scored between 0 and 100 points and a high score indicates good health status.The SF-36 scale has 8 sub-parameters including general health perception, physical function, social function, pain, mental health, role difficulties due to physical causes, role difficulties due to emotional causes and vitality and includes 11 questions with a total of 36 items.
Pain Catastrophizing Scale | 3 mounths
  This scale, developed by Sullivan et al. (1995), measures the exaggerated negative mental reaction of individuals to current or anticipated painful experiences and the extent to which they catastrophize pain.The reliability and validity of the Turkish version of the scale was demonstrated by Uğurlu et al. (2017) and consists of 13 items.Each item is scored as never=0, slightly=1, moderately=2, greatly=3 and always=4.A high total score indicates a high degree of catastrophizing of pain.
Fatigue Severity Scale | 3 mounths
  It is a scale that evaluates fatigue and consists of 9 questions. Each item is scored between 0 and 7. The total score is divided by 9 and a mean score of <4 indicates no fatigue and a mean score of ≥4 indicates fatigue.
Tampa Scale of Kinesiophobia | 3 mounths
  This scale is a 17-question scale developed to measure fear of movement/reinjury.The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities
Fibromyalgia Impact Questionnaire | 3 mounths
  It is used to evaluate the health status and physical functionality of the individual diagnosed with fibromyalgia. It is a 10-question scale that assesses physical function, work status, productivity level, depression, anxiety, sleep, pain, stiffness, fatigue and well-being.
Brief Illness Perception Questionnaire | 3 mounths
  The other 7 items in the scale have a Likert-type scoring scale from 0 to 10. The scale consists of two sub-dimensions (cognitive and emotional). The eighth item consists of an open-ended question. Individuals are asked to answer open-ended questions about the three most important reasons for the illness. A high score indicates that the illness is threatening and a low score indicates that the person is comfortable.
McGill Pain Questionnaire Short Form | 3 mounths
  Developed by Melzack in 1987 and the validity and reliability of the Turkish version has been demonstrated, the questionnaire is widely used to measure pain. This questionnaire consists of a total of 15 descriptive words to determine the sensory (11 words) and effective (4 words) characteristics of pain. In this section, pain intensity (0=absent, 1=mild, 2=moderate, 3=severe) is assessed to arrive at three pain scores (sensory, effective and total pain ratio = sensory + effective). In addition, the pain felt at the time of the measurement is calculated with the Visual Analog Scale (VAS) and the total pain intensity is calculated with a 6-point Likert scale. In this scale, 0: no pain, 1: mild, 2: uncomfortable, 3: distressing, 4: terrible, 5: unbearable pain.
Central Sensitization Scale | 3 mounths
  The Central Sensitization Scale consists of 2 parts, parts A and B. Symptoms associated with central sensitization in section A is questioned. These symptoms include sensitivity to smell, light, chemical stimuli, headache, full body pain, neck and shoulder tension, muscle stiffness and pain, skin itching/redness, depressive features, waking up restless, restless legs before sleep, sleep disturbance, low energy, anxiety attacks, impaired concentration, memory problems, worsening of symptoms with stress, frequent urge to urinate, bladder discomfort, diarrhea/constipation problems and pelvic pain. Section A contains 25 items with a total score range of 0-100. For each item in this section, one of the following responses is given: "never" (0 points), "rarely" (1 point), "sometimes" (2 points), "often" (3 points), "always" (4 points). A score of 40 and above indicates the presence of central sensitization.
  In section B, it is questioned whether the patient has been diagnosed with another.
Time Up and Go Test | 3 mounths
  The balance status of the individual is evaluated by getting up from a chair with back support, walking 3 meters at a normal walking speed and returning back to the chair and the time he/she sits on the chair is measured and recorded in seconds.The test is repeated 3 times.
6 min Walk Test | 3 mounths
  It will be used to assess the functional capacity of the patients. Patients will be asked to walk as long as possible in a 20-meter hospital corridor for 6 minutes in their own rhythm and with standard commands and the distance walked will be recorded in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat University, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No